CLINICAL TRIAL: NCT01270386
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter, Phase II Study of Apatinib as Third Line Treatment in Patients With Advanced Non-squamous and Non-small Cell Lung Cancer
Brief Title: A Study of Apatinib in Patients With Advanced Non-squamous and Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Li Zhang, Department of Medical Oncology, Cancer Center, Sun Yet Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HENGRUI 20101219
Record Dates: First submitted 2010-12-29; First posted 2011-01-05 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC; apatinib; phase II; lung; cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib (Experimental): Apatinib 750 mg qd p.o. and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib
- Placebo (Placebo Comparator): Placebo qd p.o., and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: apatinib — Apatinib 750 mg p.o. once daily
  Arms: Apatinib
Drug: placebo — placebo p.o. once daily
  Arms: Placebo

SUMMARY:
Apatinib is a tyrosin-inhibitor agent targeting at vascular endothelial growth factor receptor (VEGFR), and it's anti-angiogenesis effect has been viewed in preclinical tests. Phase I study has shown that the drug's toxicity is manageable and the maximum tolerable daily dose is 850 mg. The purpose of this study is to determine whether apatinib can improve progression free survival compared with placebo in patients with advanced non-squamous and non-small cell lung cancer who failed two lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histologically or cytologic confirmed advanced non-squamous and non-small cell lung cancer.
* At least one measurable lesion which has not received radiotherapy (larger than 10 mm in diameter by spiral CT scan)
* Have failed for 2 lines of chemotherapy including EGFR-TKI.
* ECOG performance scale 0 - 1.
* Life expectancy of more than 3 months.
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
* More than 4 weeks after operation or radiotherapy
* More than 4 weeks for cytotoxic agents or tyrosine kinase inhibitors inhibitors
* Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.25×the upper limit of normal(ULN), and serum transaminase≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN, creatinine clearance rate ≥ 50ml/min,
* signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Squamous cell carcinoma (including adenosquamous carcinoma, undifferentiated carcinoma); small cell lung cancer (including small cell and non-small cell mixed lung cancer)
* Pregnant or breastfeeding women
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Any factors that influence the usage of oral administration
* PT, APTT, TT, Fbg abnormal, Receiving the therapy of thrombolysis or anticoagulation.
* Within 4 weeks before the first use of drugs, occurs pulmonary hemorrhage (≥ CTCAE class 2) or other parts' hemorrhage (≥ CTCAE class 3).
* Long-term untreated wounds or fractures.
* Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
* Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) or low-dose aspirin (between 80mg to 100mg daily) is allowed.
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial
* Treatment with VEGFR, PDGFR, sSRC-TKI before.
* History of any second malignancies within 3 years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 8 weeks

SECONDARY OUTCOMES:
Overall Survival safety | 8 weeks
DCR(Disease control rate) | 8 weeks
ORR(objective response rate) | 8 weeks
QoL(quality of life) | 8 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Dr, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Cancer Center, Sun Yet-sen University, Guangzhou, Guangdong, China